CLINICAL TRIAL: NCT00764231
Title: A Pilot Study of a Home-based Exercise Intervention for Patients With AML
Brief Title: A Study of a Home-based Exercise Intervention for Patients With Acute Myeloid Leukaemia (AML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Toronto Rehabilitation Institute (Other)
Collaborators: University Health Network, Toronto (Other); The Leukemia and Lymphoma Society (Other)
Responsible Party: Principal Investigator, Shabbir Alibhai, Staff Physician and Senior Scientist, Toronto Rehabilitation Institute
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AML001
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Acute Myeloid Leukemia; Exercise; Fatigue; Quality of Life
Keywords: acute myeloid leukemia; exercise; fatigue; quality of life; home-based; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Motor Activity; Fatigue | interventions — Exercise; Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental): This group will undergo a 12-week home-based exercise intervention with follow-up fitness assessments.
  Interventions: Behavioral: Home-based exercise program
- Wait list control (Other): This group will go on a 12-week wait list, during which time they will be asked not to change their exercise habits. After 12 weeks, this group will participate in the exercise intervention.
  Interventions: Behavioral: Wait list

INTERVENTIONS:
Behavioral: Home-based exercise program — Subjects will be given a personalized 12-week exercise program consisting of cardiovascular, musculoskeletal and flexibility exercises by a certified exercise physiologist. They will receive fitness assessments at baseline, 6 weeks and 12 weeks.
  Other Names: exercise; fitness
  Arms: Exercise
Behavioral: Wait list — Subjects will have a 12-week waiting period, during which time they will be asked not to change their exercise habits. These subjects will receive the same fitness assessments as the experimental group (baseline, 6 weeks, 12 weeks), but will not receive an exercise program during the wait-list period. Following the 12-week wait-list period, subjects will be given the same home-based exercise intervention as the experimental group.
  Other Names: exercise; fitness
  Arms: Wait list control

SUMMARY:
Fatigue is the most common and disabling symptom in acute myeloid leukaemia (AML). Studies in other cancer patients with fatigue have shown that exercise improves both fatigue and quality of life (QOL), but there are no such studies in AML. The investigators want to conduct a pilot study of a home-based exercise program to see if this type of exercise program is feasible for AML patients, reduces fatigue, and improves QOL. What the investigators learn from this study will be essential to designing a larger, definitive randomized trial of exercise in patients with AML.

DETAILED DESCRIPTION:
Background: Fatigue is the most common and disabling symptom affecting patients with acute myeloid leukaemia (AML). Fatigue is negatively associated with quality of life (QOL) and daily function, and remains a major problem for patients even 6 months after completion of treatment (12 months after diagnosis). Despite this, there have been no intervention studies to reduce fatigue and improve QOL in AML. In a number of studies done in mostly younger patients with solid tumours, exercise has been shown to improve fatigue and QOL. Because of important differences between older patients with AML and younger patients with solid tumours, a randomized trial needs to be performed in this population. Prior to embarking on a definitive study, a pilot study is needed to ensure feasibility, to estimate recruitment rates, and to demonstrate if exercise is effective in reducing fatigue in older patients with AML.

Objectives: (1) To determine the feasibility of recruitment to, and patient adherence with, a 12-week home-based exercise intervention study among patients age 40 or older with AML in complete remission. (2) To provide estimates of the effects of exercise on fatigue and QOL to facilitate the design of a RCT. (3) To examine the relationship between exercise adherence, improvements in fitness, fatigue, and QOL in AML patients undergoing a home-based exercise intervention.

Methods: Patients age 40 or older with AML who have completed chemotherapy and achieved complete remission are eligible for the study. Patients will be recruited at the Princess Margaret Hospital, Canada's largest AML referral centre. Fitness and QOL measures will be assessed at baseline, half-way through the intervention, at the end of the 12-week exercise intervention, and 12 weeks later. Patients will be randomized to the intervention arm or a wait-list control. The intervention consists of a structured, personalized, 12-week home-based exercise program that is theory-based and modelled after a successful program in patients with another malignancy. A certified fitness instructor will lead the intervention. Patients in the wait-list control group will be asked to maintain usual level of activity for 12 weeks, after which they will be crossed over to the intervention arm to receive an identical intervention. Fitness measures include anthropometric measures, the 6-minute walk test, grip strength, and a measure of flexibility. The primary outcome measure is fatigue, which will be measured with the FACT Fatigue subscale. QOL will be assessed with the EORTC QLQ-C30. Weekly telephone assessments and 5 in-clinic assessments over the duration of the program will be done to measure program adherence. The investigators plan to approach 100 patients over a 12-month period and anticipate recruiting 40 patients. A detailed recruitment log will be maintained. Mixed effects linear regression models will be used to measure the effect of the intervention on fatigue and QOL. Relationships between changes in fitness level will be regressed with changes in fatigue and QOL in a secondary analysis. The impact of exercise adherence on outcomes will also be assessed.

Significance: Despite the importance of fatigue in patients with AML, its treatment remains poorly understood.The investigators plan to evaluate the most promising intervention, exercise, in a pilot study. The results of our study will be crucial to the design of a definitive multi-centre randomized trial to lessen fatigue and improve overall QOL in middle-aged and older patients with AML.

ELIGIBILITY:
Inclusion Criteria:

* Completion of induction and consolidation chemotherapy
* AML with histologically confirmed complete remission
* Fluency in English (or availability of bilingual caregiver and fluency in language for which validated translations of the FACT-Fatigue exist)
* Potential participants must also be screened with the Physical Activity Readiness Questionnaire (PAR-Q & PAR-MedX) and receive physician approval to participate in an exercise program

Exclusion Criteria:

* Another active malignancy
* Life expectancy < 3 months
* Severe or unstable cardiorespiratory disease
* Bone marrow transplant candidates

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-10; Primary Completion 2011-02 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Quality of life (fatigue, global health) | 12 weeks

SECONDARY OUTCOMES:
Recruitment rate | 12 weeks
Adherence rate | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shabbir MH Alibhai, MD, MSc, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada